CLINICAL TRIAL: NCT05437432
Title: Esthetic Evaluation of Onlay Restorations Constructed From Two Types of Glass Ceramics:A Randomized Clinical Trial.
Brief Title: Esthetic Evaluation of Onlay Restorations Constructed From Vita Ambria Glass Ceramics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohammed Abdelhameed, Assistant lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Color of Vita Ambria
Record Dates: First submitted 2022-06-25; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Dental Caries; Tooth Decay
Keywords: Inlay, e.max, Vita ambria, glass, cermaics, onlay, overlay
MeSH Terms: conditions — Dental Caries; Chromosome 2q32-Q33 Deletion Syndrome | interventions — IPS e.max Press

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vita ambria onlay restoration (Experimental): onlays constructed from zirconia-reinforced lithium disilicate glass ceramic press system
  Interventions: Procedure: VITA AMBRIA
- e.max onlay restoration (Active Comparator): onlays constructed from lithium disilicate glass ceramic press system
  Interventions: Procedure: IPS e.max press

INTERVENTIONS:
Procedure: VITA AMBRIA — 25 onlay restroations will be fabricated from Vita-ambria glass ceramic press system.
  Other Names: Zirconia-reinforced lithium disilicate glass ceramic press system
  Arms: Vita ambria onlay restoration
Procedure: IPS e.max press — 25 onlay restroations will be fabricated from IPS e.max glass ceramic press system.
  Other Names: Lithium disilicate glass ceramic press system
  Arms: e.max onlay restoration

SUMMARY:
There is limited data available on VITA AMBRIA glass ceramic , so this study is conducted to investigate the esthetic parameters of this new glass press system.

DETAILED DESCRIPTION:
This study will be randomized, double blinded, 1:1 parallel group, superiority clinical trial. including two research groups; VITA AMBRIA ( intervention) and IPS e.max press( Comprator). The total subjects in this study are 50, recruited from the faculty' out patient clinic. 50 partial coverage indirect restorations will fabricated and cemented for each subject. Clinical evaluations will be conducted at baseline, 6, and 12 months of follow-up according to FDI World Dental Federation criteria by two independent evaluators. The primary outcome is examining the color stability and translucency.

ELIGIBILITY:
Inclusion Criteria:

Participants in this trial should be Healthy, between 18-50 years old, have normal occlusion, well aligned teeth, and good oral hygiene. Both sexes will be included. Participants should present with one or more of their posterior teeth having moderate-size coronal decay or old filling. The target teeth should be free from any signs and symptoms and should have complete root apex with no fracture as determined by the radiograph.

Exclusion Criteria:

Incapable of self-care, mental illness, undergoing radiotherapy, epilepsy, diabetic patient, pregnancy, allergy to one of the materials used, smokers, parafunctional habits, poor oral hygiene, severe periodontitis, teeth need surgical crown lengthening or marginal elevation, teeth with enamel discoloration or enamel/dentin hypoplasia or hypocalcification, Malaligned or malformed teeth and adjacent or opposing teeth are missed. Third molars and teeth need vital pulp therapy will also be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Color stability and translucency | 12 months
  According to FDI criteria;
  1. Color and translucency of the restoration have a clinically excellent colour match with the surrounding enamel and adjacent teeth. There is no difference in shade, brightness or translucency between restoration and tooth.
  2. Colour match is clinically acceptable but minor deviations in shade between tooth and restoration are apparent.
  3. Colour match is satisfactory; there is a clear deviation in colour match that does not affect aesthetics.
  4. Colour and/or translucency are clinically unsatisfactory. There is a localized discoloration or opaqueness in the restoration making it immediately recognizable from a speaking distance and affecting the appearance of the dentition. Partial removal and repair are possible.
  5. Colour match and/or translucency. are clinically unsatisfactory. The restoration displays an unacceptable alteration in colour and/or translucency. Restoration needs replacement.

SECONDARY OUTCOMES:
Surface gloss/Luster | 12 months
  1.1 Luster comparable to enamel. 1.2.1 Slightly dull, not noticeable from speaking distance. 1.2.2 Some isolated pores. 1.3.1 Dull surface but acceptable if covered with film of saliva. 1.3.2 Multiple pores on more than one third of the surface. 1.4.1 Rough surface cannot be masked by saliva film, simple polishing is not sufficient. Further intervention necessary.
  1.4.2 Voids. 1.5 Very rough, unacceptable plaque retentive surface.
Staining a. surface b. margin | 12 months
  2a.1 No surface staining. 2b.1 No marginal staining. 2a.2 Minor surface staining, easily removable by polishing. 2b.2 Minor marginal staining, easily removable by polishing. 2a.3 Moderate surface staining that may also present on other teeth, not esthetically unacceptable.
  2b.3 Moderate marginal staining, not esthetically unacceptable. 2a.4 Unacceptable surface staining on the restoration and major intervention necessary for improvement.
  2b.4 Pronounced marginal staining; major intervention necessary for improvement.
  2a.5 Severe surface staining and/or subsurface staining, generalized or localized, not accessible for intervention.
  2b.5 Deep marginal staining, not accessible for intervention.
Esthetic anatomical form | 12 months
  4.1 Form is ideal. 4.2 Form is only slightly deviated from the normal. 4.3 Form deviates from the normal but is esthetically acceptable. 4.4. Form is affected and unacceptable esthetically. Intervention/correction is necessary.
  4.5 Form is unsatisfactory and/or lost. Repair not feasible / reasonable, Replacement needed.

CONTACTS AND LOCATIONS:
Overall Officials: Hussein R Mohamed, Study Director — Assistant Professor of Crown and Bridge Faculty of Dental Medicine, Boys, Cairo Al-Azhar University; Ahmad M El Kouedi, Study Chair — Professor of Crown and Bridge Faculty of Dental Medicine, Boys, Cairo Al-Azhar University
Locations (1):
- Faculty of Dental Medicine, Boys, Cairo Al-Azhar University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azeem RA, Sureshbabu NM. Clinical performance of direct versus indirect composite restorations in posterior teeth: A systematic review. J Conserv Dent. 2018 Jan-Feb;21(1):2-9. doi: 10.4103/JCD.JCD_213_16. PMID 29628639
- [Background] Pop-Ciutrila IS, Ghinea R, Dudea D, Ruiz-Lopez J, Perez MM, Colosi H. The effects of thickness and shade on translucency parameters of contemporary, esthetic dental ceramics. J Esthet Restor Dent. 2021 Jul;33(5):795-806. doi: 10.1111/jerd.12733. Epub 2021 Apr 18. PMID 33866673
- See also: Clinical performance of direct versus indirect composite restorations in posterior teeth: A systematic review — https://www.jcd.org.in/article.asp?issn=0972-0707;year=2018;volume=21;issue=1;spage=2;epage=9;aulast=Azeem